CLINICAL TRIAL: NCT01805934
Title: Quadruple Therapy With Furazolidone Versus Dual Therapy With High Doses of Amoxicillin as Rescue Regimens for Helicobacter Pylori Infection
Brief Title: Quadruple Therapy Versus Dual Therapy as Rescue Regimens for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Xiaobo Li, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rjyyxhk2013-01
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Rescue Therapy for Helicobacter Pylori
Keywords: Helicobacter pylori, rescue, quadruple therapy，dual therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group RBLF (Active Comparator): receive a 14-day quadruple therapy,including rabeprazole(10mg bid),bismuth citrate(220mg bid),levofloxacin(200mg qm) and furazolidone(100mg bid).
  Interventions: Drug: RBLF
- Group RA (Active Comparator): receive a 14-day dual therapy with high doses of rabeprazole(20mg bid) and amoxicillin(1000mg tid).
  Interventions: Drug: RA

INTERVENTIONS:
Drug: RBLF — The patients in Group RBLF will receive a 14-day quadruple therapy,including rabeprazole(10mg bid),bismuth citrate(220mg bid),levofloxacin(200mg qm) and furazolidone(100mg bid).
  Arms: Group RBLF
Drug: RA — The patients in Group RA will be sent to a penicillin skin test before treatment except they were given penicillin before. They will receive a 14-day dual therapy with high doses of rabeprazole(20mg bid) and amoxicillin(1000mg tid).
  Arms: Group RA

SUMMARY:
The eradication rates of first-line treatment for Helicobacter pylori(Hp) infection are not satisfactory. The study aims to compare the efficacy and safety between quadruple therapy with furazolidone and dual therapy with high doses of amoxicillin as rescue regimens for Hp.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 80 years, who presented with upper gastrointestinal symptoms and endoscopically proven H. pylori-positive non-ulcer dyspepsia, were recruited into the study.

Exclusion Criteria:

* patients with peptic ulcer,
* previous H. pylori eradication treatment,
* previous gastric surgery,
* pregnancy,
* lactation,
* major systemic diseases,
* receipt of anti-secretory therapy,
* antibiotics or bismuth in the preceding four weeks, or - allergy to any one of the medications in the regimen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
13C-urea breath test | 4 weeks after treatment
  When the outcome of 13C-urea breath test is more than 4%, the helicobacter pylori infection is still exist(positive).

SECONDARY OUTCOMES:
scale analysis of drug safety | 4 weeks after treatment

OTHER OUTCOMES:
13C-urea breath test | baseline

CONTACTS AND LOCATIONS:
Overall Officials: xiaobo Li, MD, Study Director — RenJi Hospital
Locations (1):
- Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China